CLINICAL TRIAL: NCT02922803
Title: Vitamin D and Physical Performance Before and After Intervention and Birth Outcome in Pregnant Somali and Swedish Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Paul Kalliokoski, MD, Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DVITOS2
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Muscle Weakness; Vitamin D Deficiency
MeSH Terms: conditions — Muscle Weakness; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D insufficient (Active Comparator): Subjects with Vitamin D level in blood > 25 nmool/L < 50 nmol/L will be treated with 1 combination tablet of Vitamin D3/calcium per day
  Interventions: Drug: 1 combination tablet of Vitamin D3/calcium per day
- Vitamin D deficient (Active Comparator): Subjects with Vitamin D level in blood < 25 nmol/L (25-OHD) will be treated with 2 combination tablets of Vitamin D3/calcium per day
  Interventions: Drug: 2 combination tablets of Vitamin D3/calcium per day

INTERVENTIONS:
Drug: 1 combination tablet of Vitamin D3/calcium per day — Combination tablet of Cholecalciferol (800 IU or 20 ug) and calcium carbonate (500 mg)
  Other Names: 1 tablet Kalcipos D Forte
  Arms: Vitamin D insufficient
Drug: 2 combination tablets of Vitamin D3/calcium per day — Combination tablets of Cholecalciferol (800 IU or 20 ug) and calcium carbonate (500 mg)
  Other Names: 2 tablets Kalcipos D Forte
  Arms: Vitamin D deficient

SUMMARY:
Somali migrant women, often in veiled clothing, living in a town in mid Sweden on the 60:th parallel were observed to be weak and to have a waddling gate.

Study 1 was carried out in the setting of an antenatal clinic administered from a primary care center in Borlänge, a Swedish middle-sized industrial town at the 60:th parallel in Sweden. The investigators chose an initial study period in late spring to reflect the effects of the dark season with little ultraviolet B radiation that affects vitamin D production. Study 1 was carried out in a short period of time. The recruitment was performed in a retrospective design in order to neglect the seasonal effects of ultraviolet B radiation. Study 1 was carried out in year 2010. It was a cross sectional baseline study of blood levels of vitamin D measured as 25-hydroxyvitamin D (25-OHD) and physical performance in 123 pregnant and new mothers from Somalia (n=52) and Sweden (n=71).

Study 2: Examines the results on muscular performance, i.e. grip strength and squatting ability, from intervention with advice and prescription of vitamin D3 and calcium for 10 months, in all the women from study 1 with 25-OHD levels <50 nmol/L or 50 nmol/L of 25-OHD.

Study 3: The recruitment to Study 1 also serves as recruitment for a cohort study on delivery outcome in birth protocols starting 2016.

Study 4: The aim is to study the emic perspective and lifestyle related to vitamin D and strength in the group of Somali women by focus interviews among the Somali women from above.

A possible fifth study will explore correlations between 25-OHD and pain distribution and pain parameters.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or new mother from Sweden or Somalia living in Borlänge and registered the antenatal clinic in Borlänge maximally 21 months prior to study start.

Exclusion Criteria:

* Severe metabolic, medical or mental disease (ex. deranged type I diabetes or psychosis).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2010-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
S-25-hydroxyvitamin D in nmol/L. | 10 months
Grip strength in Newton. | 10 months
Upper leg strength, able or not able to squat | 10 months

SECONDARY OUTCOMES:
Trendelenburg's sign positive or not. not. | 10 months
Sit to stand five times, able or not. | 10 months
Standing on one leg 30 seconds, able or not | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kalliokoski, MD, Principal Investigator — Uppsala University; Monica Löfvander, Ass. Prof., Study Director — Uppsala University
Locations (1):
- Primary Health care center Jakobsgårdarna, Borlänge, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalliokoski P, Bergqvist Y, Lofvander M. Physical performance and 25-hydroxyvitamin D: a cross-sectional study of pregnant Swedish and Somali immigrant women and new mothers. BMC Pregnancy Childbirth. 2013 Dec 17;13:237. doi: 10.1186/1471-2393-13-237. PMID 24345271
- [Derived] Kalliokoski P, Widarsson M, Rodhe N, Lofvander M. Positive impact on vitamin D related lifestyle of medical advice in pregnant Somali-born women and new mothers: a mixed method study in Swedish primary care. BMC Public Health. 2021 Feb 5;21(1):297. doi: 10.1186/s12889-021-10277-y. PMID 33546641
- [Derived] Kalliokoski P, Rodhe N, Bergqvist Y, Lofvander M. Long-term adherence and effects on grip strength and upper leg performance of prescribed supplemental vitamin D in pregnant and recently pregnant women of Somali and Swedish birth with 25-hydroxyvitamin D deficiency: a before-and-after treatment study. BMC Pregnancy Childbirth. 2016 Nov 15;16(1):353. doi: 10.1186/s12884-016-1117-3. PMID 27846821